CLINICAL TRIAL: NCT07362745
Title: Single-Cell and Spatial Transcriptomics Analysis of Steatotic Donor Liver Susceptibility to Post-Transplant Injury
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Wang Lin, Professor, Xijing Hospital
Other Study IDs: KY20252571-C-1
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Fatty Liver; Liver Transplant; Complications; Ischaemia Reperfusion Injury of Liver; End Stage Liver Disease; Liver Failure; Postoperative Complications
MeSH Terms: conditions — Fatty Liver; End Stage Liver Disease; Liver Failure; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steatotic Donor Liver Recipients: Liver transplant recipients receiving donor livers with macrovesicular steatosis ≥5% (steatotic donor liver). Participants undergo standard liver transplantation with two small liver tissue samples collected during surgery (during graft preparation and before abdominal closure) followed by postoperative monitoring.
- Normal Donor Liver Recipients: Liver transplant recipients receiving donor livers with <5% steatosis (normal donor liver). Participants undergo standard liver transplantation with two small liver tissue samples collected during surgery (during graft preparation and before abdominal closure) followed by postoperative monitoring.

SUMMARY:
The goal of this observational study is to understand why liver transplants from donors with fatty liver disease (steatotic donor livers) are more vulnerable to post-transplant injury, analyzing historical clinical data and collected tissue samples using advanced genetic techniques.

The main questions it aims to answer are:

* Which specific cell types and their spatial interactions contribute to increased post-transplant injury susceptibility in steatotic donor livers?
* What are the key molecular differences in gene expression between steatotic and normal donor livers following transplantation?

Researchers will compare 300 historical liver transplant cases from 2015-2025, including 50 cases with archived tissue samples available for molecular analysis, and 250 cases with clinical data only. Donor liver steatosis was assessed by histopathology when tissue was available, or by donor clinical data when tissue was not available. The two groups (steatotic donor liver recipients vs. normal donor liver recipients) will be matched based on donor age, ischemia time, recipient scores, and other key clinical parameters to control for potential confounding variables.

This is a retrospective analysis of existing data and archived biospecimens; no prospective participant enrollment or additional sample collection will occur.

ELIGIBILITY:
Inclusion Criteria:

Recipient Criteria:

* Participant (or legal representative if unable to read/sign) provides written informed consent
* Age 18-80 years (inclusive) at time of enrollment
* Clinical diagnosis of liver failure requiring liver transplantation
* Stable vital signs and deemed medically fit to tolerate liver transplantation surgery

Donor Criteria:

* Fatty degeneration range: Macrovesicular steatosis 0-30%
* Donor age: ≤60 years
* Cold ischemia time (CIT): ≤12 hours for deceased donors
* Liver function: ALT/AST <5 times upper limit of normal

Exclusion Criteria:

Recipient Criteria:

* Pregnant or lactating women
* Prior history of non-autologous (allogeneic) bone marrow or stem cell transplantation
* Blood transfusion within 7 days prior to tissue sampling
* Radical cancer treatment within 3 years prior to enrollment
* Use of anti-tumor medications within 30 days prior to enrollment
* Known bleeding diathesis or coagulation disorder
* Active autoimmune disease
* Concurrent malignancy or multiple primary tumors

Donor Criteria:

* Fibrosis: Any degree of hepatic fibrosis
* Steatohepatitis: Presence of lobular inflammation or hepatocyte ballooning
* Active infection: HBV, HCV, or HIV positive
* Severe fatty liver-related comorbidities: Uncontrolled diabetes (HbA1c>8%), severe hyperlipidemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective, single-center observational cohort study will enroll 300 adult liver transplant recipients at the First Affiliated Hospital of Air Force Medical University. The study population consists of patients aged 18-80 years with end-stage liver disease requiring orthotopic liver transplantation. Participants will be naturally grouped based on donor liver characteristics into: (1) steatotic donor liver recipients (donor livers with macrovesicular steatosis ≥5%), and (2) normal donor liver recipients (donor livers with steatosis <5%). All participants must have stable vital signs and be medically fit to tolerate liver transplantation surgery. The two groups (steatotic donor liver recipients vs. normal donor liver recipients) will be matched based on donor age, ischemia time, recipient scores, and other key clinical parameters to control for potential confounding variables.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Differential Expression of Post-Transplant Injury-Related Genes | Tissue collection at two intraoperative time points (during graft preparation and before abdominal closure); sequencing and data analysis completed within 1 year of data collection
  Quantification of injury-related gene expression changes associated with post-transplant liver injury in liver tissue samples analyzed by single-cell RNA sequencing. Expression levels will be compared between recipients of steatotic donor livers (≥5% macrovesicular steatosis) and recipients of normal donor livers (<5% steatosis) to identify molecular mechanisms underlying increased injury susceptibility.
Postoperative Liver Function Recovery and Clinical Outcomes | Up to 10 years post-transplantation, determined by retrospective data availability
  Comparison of post-transplant clinical parameters between recipients of steatotic versus normal donor livers, including serial measurements of alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and other standard liver function tests, as well as vital signs and clinical assessment data collected during postoperative follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobiliary Surgery, Xijing Hospital, Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
**Plan to Share IPD (Individual Participant Data): No**
  **Rationale:** This study involves highly sensitive personal data including genomic/transcriptomic information (single-cell and spatial transcriptomics) and detailed clinical records from human transplant recipients. Due to privacy protection requirements, Chinese regulations on human genetic data, and the need for explicit participant consent for data sharing beyond the original research purpose, individual participant data will not be shared publicly. Aggregated, de-identified results will be published in scientific reports.